CLINICAL TRIAL: NCT00865826
Title: Sensitivity and Specificity of Mycobacterium Tuberculosis Screening and Diagnostics in HIV-Infected Individuals
Brief Title: Observational Study of Specificity of Mycobacterium Tuberculosis Screening and Diagnostics in HIV-Infected Individuals
Status: Completed | Type: Observational
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACTG A5253; 1U01AI068636 (NIH)
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Pulmonary Tuberculosis; Myobacterium Infections
MeSH Terms: conditions — HIV Infections; Tuberculosis; Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum samples and blood collection

GROUPS / COHORTS (1):
- 1: HIV-infected males and females who are not currently receiving ART
  Interventions: Other: Standardized diagnostic evaluation

INTERVENTIONS:
Other: Standardized diagnostic evaluation — Participants will undergo a diagnostic evaluation for TB at study entry
  Other Names: SDE

SUMMARY:
An estimated 3 million HIV-infected individuals will enter programs for antiretroviral (ARV) treatment in the coming year, with projected rates of requirement for ARV therapy extending to more than 10 million in sub-Saharan Africa, southeastern Asia, and Latin America in the coming decade. In these settings, Tuberculosis (TB) is an endemic infection in the population, and an estimated 30-60% of adults have been infected with TB, the leading opportunistic infection associated with HIV infection. The purpose of this study is to construct a standardized diagnostic evaluation (SDE) for TB that provides an increase in identification of participants with active pulmonary TB, without sacrificing specificity.

DETAILED DESCRIPTION:
Well developed TB diagnostic testing, contact tracing, and treatment programs are key parts of the public health and health care infrastructure in many countries where HIV infection has resulted in a 3- to 10-fold increase in clinical TB, accompanied by increasing HIV prevalence. The primary purpose of this study is to construct a standardized diagnostic evaluation (SDE) for TB that provides an increase in identification of participants with active pulmonary TB, without sacrificing specificity.

This observational study will include participants who are HIV-infected and TB-uninfected and not receiving ARV therapy. The duration of this trial will last between 1 and 14 days. Screening and study entry may occur at the same visit. All evaluations must be performed within 14 days after the participant is registered. Medical and medication history, physical exam, oral examination and swab, chest x-ray, sputum and blood collection, and documentation of PPD/TST (if available) will occur within this 14-day period.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected

Exclusion Criteria:

* Receipt of ART within 90 days prior to study entry
* Diagnosis of active TB (pulmonary or extrapulmonary) within 90 days prior to study entry
* Receipt of 7 or more cumulative days of certain medications within 90 days prior to study entry. More information on this criterion can be found in the protocol.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV-infected males and females who are not currently receiving ART
Sampling Method: Probability Sample
Enrollment: 801 (Actual)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Effectiveness in creating a standard diagnostic evaluation for identification of participants with active pulmonary TB | Throughout study

SECONDARY OUTCOMES:
Prevalence of TB in symptomatic and asymptomatic individuals | Throughout study
Rates of TB drug resistance | Throughout study
Feasibility and incremental benefits of diagnostic and screening evaluations over a range of CD4 cell counts | Throughout study
Value of oral candidiasis as a predictor of TB | Throughout study
Significance of investigational serologic assay when added to sputum acid-fast bacilli (AFB) smears when identifying participants with active TB compared to AFB smears alone | Throughout study
Storage of samples for future diagnostic and pathogenesis studies of mycobacterial, virologic, and immunologic factors | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Susan Swindells, MBBS, Study Chair — University of Nebraska; Srikanth Tripathy, MBBS, Study Chair — National AIDS Research Institute, MIDC, Bhosari
Locations (13):
- Botswana (2):
  - Gaborone Prevention/Treatment Trials CRS, Gaborone
  - Molepolole Prevention/Treatment Trials CRS (Molepolole PTT CRS), Molepolole
- Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Manguinhos, Rio de Janeiro, Brazil
- India (2):
  - BJ Medical College CRS, Pune, Maharashtra
  - NARI Pune CRS, Pune, Maharashtra
- University of North Carolina Lilongwe CRS, Lilongwe, Malawi
- Peru (2):
  - San Miguel CRS, San Miguel, Lima region
  - Asociacion Civil Impacta Salud y Educacion - Miraflores, CRS, Lima
- South Africa (4):
  - Soweto ACTG CRS, Johannesburg, Gauteng
  - Wits HIV CRS, Johannesburg, Gauteng
  - CAPRISA eThekwini CRS, Durban, KwaZulu-Natal
  - Durban Adult HIV CRS, Durban, KwaZulu-Natal
- UZ-Parirenyatwa CRS (30313), Harare, Zimbabwe

REFERENCES:
- [Background] Aichelburg MC, Rieger A, Breitenecker F, Pfistershammer K, Tittes J, Eltz S, Aichelburg AC, Stingl G, Makristathis A, Kohrgruber N. Detection and prediction of active tuberculosis disease by a whole-blood interferon-gamma release assay in HIV-1-infected individuals. Clin Infect Dis. 2009 Apr 1;48(7):954-62. doi: 10.1086/597351. PMID 19245343
- [Background] Ani AE. Advances in the laboratory diagnosis of Mycobacterium tuberculosis. Ann Afr Med. 2008 Jun;7(2):57-61. doi: 10.4103/1596-3519.55680. PMID 19143160